CLINICAL TRIAL: NCT03103243
Title: A Pilot Study to Investigate a Contemplation-Based Intervention and Health Outcomes in Systemic Lupus Erythematosus Patients
Brief Title: Pilot Study to Investigate Contemplative Intervention in Lupus Patients
Acronym: LUPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Lupus Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19671
Record Dates: First submitted 2017-03-22; First posted 2017-04-06 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Lupus; SLE; Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): This is a single arm trial. All participants will be administered two baseline fMRIs and blood analysis prior to participation in a mindfulness group and individual mindfulness intervention sessions. A post intervention fMRI and blood analysis will complete the trial participation.
  Interventions: Behavioral: Mindfulness Based Group Sessions

INTERVENTIONS:
Behavioral: Mindfulness Based Group Sessions — In-person group intervention sessions conducted with a combination of meditation, group exercise (yoga), group discussions, deep breathing and other mindfulness based practices.

SUMMARY:
The study tests whether contemplative-based intervention can modify pathogenic processes in participants with Lupus. Techniques such as meditation, mindfulness and yoga may have an impact on the disease and may decrease psychological distress, increase self-regulation capabilities, and reduce pain. Additionally, incorporating patients' caregivers may strengthen their relationships and, thereby, improve their health and well-being.

DETAILED DESCRIPTION:
The objective of this pilot study is to test the feasibility of an innovative contemplative-based and caregiver-inclusive intervention can modify pathogenic processes in systemic lupus erythematosus (SLE). Contemplative techniques such as meditation, mindfulness and yoga may have an impact on the disease burden and may decrease psychological distress, increase self-regulation capabilities, and reduce pain. Research also suggests that contemplative practices, such as an intensive mindfulness intervention, may have a direct effect on the underlying disease process itself by altering epigenetic control of gene expression, decreasing proinflammatory cytokine production and reestablishing immunologic homeostasis. It is also well documented that social relationships moderate physical health. Incorporating patients' caregivers may strengthen their relationships and thereby improve their health and well-being. It is anticipated that the successful outcome of the intervention described in this proposal will provide the basis for a new and effective contemplative-based and caregiver-inclusive therapy for SLE and other rheumatic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who have given written informed consent
* 18 and older
* Literate in English: able to read, understand, follow instructions, and complete the rating scales and questionnaires accurately
* Have a clinical diagnosis of systemic lupus erythematosus
* Must pass the initial MRI screening administered over the phone
* Inclusion criteria for support person: must be able to attend sessions with SLE patient.

Exclusion Criteria:

* Significant previous mindfulness training and experience (e.g. MBSR course, daily meditation practice)
* Any current Axis I DSM-IV-TR psychiatric disorder that, in the clinician's opinion, warrants treatment or would preclude safe participation in the protocol, including, but not limited to: psychosis, schizophrenia, dementia, schizotypal personality disorder, borderline personality disorder, bipolar disorder, primary diagnosis of eating disorder, or chronic suicidality or homicidality.
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseases not related to SLE (i.e., diabetes, cardiovascular, pulmonary, hematologic, gastrointestinal, neurological, or infectious) which, in the opinion of the treating physician, could confound the results of the study or put the patients at undue risk
* Chronic use of prescribed or recreational psychoactive drugs (self-reported)
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 364 days prior to Baseline (self-reported)
* Diagnosis of lupus for over 20 years
* Too sick to meaningfully participate (e.g. hospitalized, flaring at the time of screening)
* In order to participate in the MRI portion of the study, participants must pass the in-person MRI screening administered by the MRI technician before each MRI. If participants fail the in-person MRI screening, they will be excluded from the MRI portion of the study, but can still participate in the intervention and blood draw portions of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood | Baseline Assessment, within 2 weeks prior to intervention, within 2 weeks after intervention
  Number of participants with abnormal lab values (Complete Blood Count, Chemistry Panel, Autoantibodies, Complement C3 & C4, Cytokines)

SECONDARY OUTCOMES:
Change from baseline in brain activity during functional MRI | Baseline Assessment, within 2 weeks prior to intervention, within 2 weeks after intervention
  Number of participants with change in brain activity during functional MRI tasks (Handholding, Balloon Analog Risk Task, Penn Emotion Recognition Task, Operation Span Task, Resting State Task)
Change from baseline in Patient Reported Outcomes | Baseline Assessment, within 2 weeks prior to intervention, throughout the 6-week intervention, within 2 weeks after intervention
  Patient-reported change in health and symptoms
Change from baseline in SLE disease activity | Baseline Assessment, within 2 weeks prior to intervention, within 2 weeks after intervention
  Systemic Lupus Activity Questionnaire (SLAQ)
Change from baseline in psychosocial function | Baseline Assessment, within 2 weeks prior to intervention, throughout the 6-week intervention, within 2 weeks after intervention
  Self reported psychosocial function
Change from baseline in Heart Rate Variability | Throughout the entire 6-week intervention
  Collected using emWave device

CONTACTS AND LOCATIONS:
Overall Officials: James A Coan, Ph.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No